CLINICAL TRIAL: NCT01099241
Title: Use of Ultrasound to Determine Central Venous Pressure in Critically Ill Patients
Brief Title: Central Venous Pressure (CVP) Assessment by Ultrasound and Physical Examination
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Gregory A. Schmidt, MD, Roy J. & Lucille A. Carver College of Medicine, University of Iowa
Other Study IDs: 20076777
Record Dates: First submitted 2010-03-26; First posted 2010-04-06 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-03

CONDITIONS: Central Venous Pressure
Keywords: CVP; US; Ultrasonography

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ultrasound may be useful for noninvasively determining the central venous pressure. We intend to compare the clinical examination of the neck veins; ultrasound delineation of the internal jugular vein; and the central venous pressure measured with an intravascular catheter.

ELIGIBILITY:
Inclusion Criteria:

* adult medical or surgical ICU patients who have preexisting central venous (jugular/subclavian only) catheters.

Exclusion Criteria:

* subjects with only a femoral venous catheter.
* subjects whose CVP measurement by the indwelling catheter exceeds 20cm of water.
* subjects younger than 18 years old.
* inability to obtain informed consent from the subject or the subjects authorized representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Correlation of CVP measurement via ultrasound and central venous catheter | At data collection: this is a physiologic study
  CVP as determined non-invasively with the transcutaneous ultrasound probe will correlate with a high degree of accuracy to the measurement obtained invasively by the catheter and pressure transducer.

SECONDARY OUTCOMES:
Correlation of CVP measurement via physical examination of IJV and EJV. | At data collection: physiologic study
  Despite its more tortuous course and smaller caliber, the external jugular vein will be as reliable (compared to the catheter) as the internal jugular to estimate CVP

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Schmidt, Principal Investigator — Roy J. & Lucille A. Carver College of Medicine, University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Baumann UA, Marquis C, Stoupis C, Willenberg TA, Takala J, Jakob SM. Estimation of central venous pressure by ultrasound. Resuscitation. 2005 Feb;64(2):193-9. doi: 10.1016/j.resuscitation.2004.08.015. PMID 15680529
- [Background] Bazaral M, Harlan S. Ultrasonographic anatomy of the internal jugular vein relevant to percutaneous cannulation. Crit Care Med. 1981 Apr;9(4):307-10. doi: 10.1097/00003246-198104000-00004. PMID 7214938
- [Background] Cook DJ. Clinical assessment of central venous pressure in the critically ill. Am J Med Sci. 1990 Mar;299(3):175-8. doi: 10.1097/00000441-199003000-00006. PMID 2316561
- [Background] Davison R, Cannon R. Estimation of central venous pressure by examination of jugular veins. Am Heart J. 1974 Mar;87(3):279-82. doi: 10.1016/0002-8703(74)90064-7. No abstract available. PMID 4812363
- [Background] Lipton B. Estimation of central venous pressure by ultrasound of the internal jugular vein. Am J Emerg Med. 2000 Jul;18(4):432-4. doi: 10.1053/ajem.2000.7335. PMID 10919533
- [Background] Lipton BM. Determination of elevated jugular venous pressure by real-time ultrasound. Ann Emerg Med. 1999 Jul;34(1):115. doi: 10.1016/s0196-0644(99)70287-8. No abstract available. PMID 10409088
- [Background] Rizvi K, Deboisblanc BP, Truwit JD, Dhillon G, Arroliga A, Fuchs BD, Guntupalli KK, Hite D, Hayden D; NIH/NHLBI ARDS Clinical Trials Network. Effect of airway pressure display on interobserver agreement in the assessment of vascular pressures in patients with acute lung injury and acute respiratory distress syndrome. Crit Care Med. 2005 Jan;33(1):98-103; discussion 243-4. doi: 10.1097/01.ccm.0000150650.70142.e9. PMID 15644654
- [Background] Vinayak AG, Levitt J, Gehlbach B, Pohlman AS, Hall JB, Kress JP. Usefulness of the external jugular vein examination in detecting abnormal central venous pressure in critically ill patients. Arch Intern Med. 2006 Oct 23;166(19):2132-7. doi: 10.1001/archinte.166.19.2132. PMID 17060544
- [Derived] Deol GR, Collett N, Ashby A, Schmidt GA. Ultrasound accurately reflects the jugular venous examination but underestimates central venous pressure. Chest. 2011 Jan;139(1):95-100. doi: 10.1378/chest.10-1301. Epub 2010 Aug 26. PMID 20798190